CLINICAL TRIAL: NCT00315237
Title: Prospective, Randomized Phase III Trial of I.V. Vinflunine Plus Best Supportive Care as Second Line Therapy Versus Best Supportive Care After a Platinum-containing Regimen, in Patients With Advanced Transitional Cell Carcinoma of Urothelial Tract
Brief Title: Phase III Trial of Vinflunine Plus Best Supportive Care vs. Best Supportive Care in Patients With Transitional Cell Carcinoma (TCC) of the Urothelial Tract
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Organization: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L0070 IN 302 P1; CA183004
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Transitional Cell Carcinoma of the Urothelial Tract; Bladder Cancer; Bladder Neoplasms
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: vinflunine and best supportive care
- 2 (No Intervention): best supportive care for 18 week duration

INTERVENTIONS:
Drug: vinflunine and best supportive care — solution for injection, IV, 280/320 mg/m2, every 3 wks variable duration
  Arms: 1

SUMMARY:
The purpose of this clinical research study is to learn if patients who receive vinflunine plus best supportive care live longer than patients who receive best supportive care alone. This study will also investigate patient benefit, safety and whether or not vinflunine shrinks or slows the growth of the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer
* Progressed after 1st line platinum-chemotherapy
* >= 18 years old
* Adequate hematologic, hepatic & renal function

Exclusion Criteria:

* CNS disease
* Moderate neuropathy
* More than 1 previous chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
duration of Overall Survival after Randomization | 30-March-07

SECONDARY OUTCOMES:
patient benefit | 30-Mar-07
safety | 30-Mar-2007
response rate | throughout the study
time to response | upon occurrence
response duration | throughout the study
progression free survival | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- Canada (10):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Brampton, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, Kingston, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec

REFERENCES:
- [Derived] Rassy EE, Bakouny Z, Aoun F, Haddad FG, Sleilaty G, Assi T, Kattan J. A network meta-analysis of the PD(L)-1 inhibitors in the salvage treatment of urothelial bladder cancer. Immunotherapy. 2018 Jun;10(8):657-663. doi: 10.2217/imt-2017-0190. Epub 2018 Mar 22. PMID 29562804